CLINICAL TRIAL: NCT00088582
Title: A Multicenter, Randomized, Crossover, Open Label Dose Finding Study to Compare the Safety, Efficacy and PK/PD Relationship of Multiple Doses of SOM230 and Sandostatin in Acromegalic Patients
Brief Title: Study Comparing SOM230 Subcutaneously and Sandostatin Subcutaneously in Acromegalic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2201
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Acromegaly
Keywords: Acromegaly; SOM230; Sandostatin
MeSH Terms: conditions — Acromegaly | interventions — pasireotide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sandostatin s.c. (Octreotide) (Experimental)
  Interventions: Drug: Pasireotide (SOM230), Octreotide (Sandostatin)
- Pasireotide (SOM230) (Experimental)
  Interventions: Drug: Pasireotide (SOM230), Octreotide (Sandostatin)

INTERVENTIONS:
Drug: Pasireotide (SOM230), Octreotide (Sandostatin)

SUMMARY:
5 month study comparing SOM230 s.c. and Sandostatin s.c. in acromegalic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active acromegaly due to a pituitary adenoma
* Patients who have been previously treated for acromegaly with certain medications may be required to be without certain medications prior to entering the study

Exclusion Criteria:

* Patients with compression of the optic chiasm causing any visual field defect
* Patients who require a surgical intervention for relief of any sign or symptom associated with tumor compression
* Patients who have received radiotherapy in the 2 years prior to the start of the trial
* Patients who have congestive heart failure, unstable angina, cardia arrhythmia, or a history of acute myocardial infarction within the three months preceding enrollment
* Patients with gallstone disease
* Patients with chronic liver disease
* Known hypersensitivity to Sandostatin or Sandostatin LAR
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control and highly effective method for birth control
* History of immunocompromise, including a positive HIV test result
* Patients who have a history of alcohol or drug abuse in the six-month period prior to the enrollment visit
* Patients who have participated in any clinical investigation with an investigational drug within 4 weeks prior to dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-03; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Circulating GH- and IGF-1 concentrations measured every 2 weeks | 6 months

SECONDARY OUTCOMES:
Safety and efficacy of multiple doses of Pasireotide s.c. and Sandostatin s.c. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - New York University/VA Medical Center, New York, New York
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Result] Petersenn S, Schopohl J, Barkan A, Mohideen P, Colao A, Abs R, Buchelt A, Ho YY, Hu K, Farrall AJ, Melmed S, Biller BM; Pasireotide Acromegaly Study Group. Pasireotide (SOM230) demonstrates efficacy and safety in patients with acromegaly: a randomized, multicenter, phase II trial. J Clin Endocrinol Metab. 2010 Jun;95(6):2781-9. doi: 10.1210/jc.2009-2272. Epub 2010 Apr 21. PMID 20410233